CLINICAL TRIAL: NCT02048618
Title: Double-Blind, Randomized, Placebo-Controlled, Multi-Centre Study to Investigate the Efficacy and Safety of GLPG0634 in Subjects With Active Crohn's Disease With Evidence of Mucosal Ulceration
Brief Title: Efficacy and Safety of GLPG0634 in Subjects With Active Crohn's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Galapagos NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GLPG0634-CL-211; 2013-002857-32 (EudraCT Number)
Record Dates: First submitted 2014-01-27; First posted 2014-01-29 (Estimated); Last update posted 2016-02-23 (Estimated); Status verified 2016-02

CONDITIONS: Crohn's Disease
Keywords: Active Crohn's Disease; GLPG0634
MeSH Terms: conditions — Crohn Disease | interventions — GLPG0634

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- GLPG0634 200 mg QD (Experimental): 2 tablets of 100 mg GLPG0634 in the morning
  Interventions: Drug: GLPG0634
- GLPG0634 100 mg QD (Experimental): 1 tablet of 100 mg GLPG0634 and 1 placebo tablet in the morning
  Interventions: Drug: GLPG0634; Drug: Placebo
- Placebo QD (Placebo Comparator): 2 placebo tablets in the morning
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GLPG0634 — 100 mg oral tablet, intake once daily for 20 weeks
  Other Names: GLPG0634 tablets
  Arms: GLPG0634 100 mg QD; GLPG0634 200 mg QD
Drug: Placebo — placebo oral tablets, intake once daily for 20 weeks
  Other Names: Placebo tablets
  Arms: GLPG0634 100 mg QD; Placebo QD

SUMMARY:
* 180 patients suffering from active Crohn's disease with evidence of mucosal ulceration will be evaluated for improvement of disease activity (efficacy) when taking GLPG0634 or matching placebo once daily for 20 weeks in addition to their stable background treatment.
* During the course of the study, patients will also be examined for any side effects that may occur (safety and tolerability), and the amount of GLPG0634 present in the blood (Pharmacokinetics) as well as the effects of GLPG0634 on disease- and mechanism of action-related parameters in the blood and stool (Pharmacodynamics) will be determined. Also, the effects GLPG0634 administration on subjects' quality of life will be evaluated.

DETAILED DESCRIPTION:
* 180 patients suffering from active Crohn's disease with evidence of mucosal ulceration will be evaluated when taking GLPG0634 or matching placebo once daily in addition to their stable background treatment. The population will include 50% anti-TNF naïve patients and 50% of subjects previously exposed to anti-TNF.
* The study will consist of 2 parts, with total treatment duration of 20 weeks. Randomisation in Part 1 will be stratified according to subject's previous anti-TNF exposure, C-reactive protein (CRP) level at Screening and oral corticosteroid use at Day -1. However, at Week 10, subjects will be re-randomized automatically and stratified according to the subject's clinical response (reduction of Crohn's Disease Activity Index (CDAI) of 100 points), previous anti-TNF exposure and corticosteroid use at Day -1 to receive GLPG0634 200 mg q.d., 100 mg q.d. doses, or matching placebo q.d. in a blinded fashion. In Part 2, all will continue the study until Week 20.
* As efficacy parameters, the ability to achieve clinical response or remission, endoscopic response & remission as well as mucosal healing with GLPG0634 given once daily compared to placebo will be evaluated after 10 weeks of treatment. In subjects who achieved clinical remission at Week 10, maintenance of the remission will be assessed during Part 2 of the study.
* During the course of the study, patients will also be examined for any side effects that may occur (safety and tolerability), and the amount of GLPG0634 present in the blood (Pharmacokinetics) as well as the effects of GLPG0634 on disease- and mechanism of action-related parameters in the blood and stool (Pharmacodynamics) will be determined. Also, the effects of different doses and dose regimens of GLPG0634 administration on subjects' quality of life will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects between 18 and 75 years
* Documented history of ileal, colonic, or ileocolonic CD
* CDAI score ≥ 220 to ≤ 450
* Evidence of active inflammation as demonstrated by endoscopic confirmation of active disease
* Subjects previously not exposed to anti-TNF treatment (TNF-naïve) or subjects previously exposed to anti-TNF therapy at a registered dose, that has been discontinued at least 8 weeks prior to Screening and deemed by the treating physician as a primary or secondary non-responder or intolerant (TNF-experienced)
* Continuation of concurrent treatment with oral steroids (≤30 mg prednisolone eq/day), mesalazine, olsalazine, CD-related antibiotics and probiotics at stable dose is allowed
* Previous exposure to immunomodulators is permitted, but must be discontinued
* Haematology and biochemistry lab parameters within predefined ranges as stated in the protocol

Exclusion Criteria:

* Diagnosis of indeterminate colitis, ulcerative colitis (UC), or clinical findings suggestive of UC
* Stoma, gastric or ileoanal pouch, procto- or total colectomy, symptomatic stenosis or obstructive strictures, history of bowel perforation, (suspected) abscess; actively draining fistulae
* Subject who has had surgical bowel resections within the past 6 months, short bowel syndrome or is receiving tube feeding, defined formula diets, or parenteral alimentation
* Subject with positive Clostridium difficile toxin stool assay or evidence of any other gastrointestinal infection
* Subject who has received non-permitted IBD therapies within specified timeframes, depending on the medication, as stated in the protocol
* Subject with a (previous history of) dysplasia of the gastrointestinal tract
* Concurrent gastro-intestinal malignancy or a history of cancer elsewhere
* History of lymphoproliferative disease
* Known active infection of any kind, current therapy for chronic infection or history of specific infections as stated in the protocol
* Subject who is pregnant, lactating or not willing to maintain highly effective birth control methods during the course of the study and 12 weeks thereafter

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2014-02; Primary Completion 2015-11 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects achieving clinical remission at Week 10 | Week 10
  Percentage of subjects achieving clinical remission as defined by a Crohn's Disease Activity Index score < 150 points

SECONDARY OUTCOMES:
Percentage of subjects achieving clinical remission | Up to Week 20
  Percentage of subjects achieving clinical remission as defined by a Crohn's Disease Activity Index score < 150 points, assessed at every visit
Percentage of subjects achieving clinical response | Up to Week 20
  Percentage of subjects achieving clinical response as defined by a decrease in Crohn's Disease Activity Index score of at least 100 points, assessed at every visit
Percentage of subjects achieving endoscopic remission at Week 10 | Week 10
  Percentage of subjects achieving endoscopic remission as defined by a reduction of Simplified Endoscopy Score for Crohn's Disease (SES-CD) score ≤ 4, with ulcerated surface subscore no greater than 1 in any segment at Week 10
Percentage of subjects achieving endoscopic response at Week 10 | Week 10
  Percentage of subjects achieving endoscopic response as defined by a reduction of Simplified Endoscopy Score for Crohn's Disease (SES-CD) score by at least 50% from Screening at Week 10
Percentage of subjects achieving mucosal healing at Week 10 | Week 10
  Percentage of subjects achieving mucosal healing as defined by a Simplified Endoscopy Score for Crohn's Disease (SES-CD) score equal to 0 at Week 10
Change from Baseline in Crohn's Disease Activity Index score | Up to Week 20
  Change from Baseline in Crohn's Disease Activity Index score, assessed at every visit
Change from Screening in endoscopic score | Week 10
  Change from Screening in endoscopic Simplified Endoscopy Score for Crohn's Disease (SES-CD) score at Week 10
Change from Screening in histopathology biopsy score | Week 10
  Change from Screening in histopathology biopsy score at Week 10
Change from Baseline in Subjects' Quality of Life (based on the Inflammatory Bowel Disease Questionnaire (IBDQ) questionnaire score) | Up to Week 20
  Change from Baseline in Subjects' Quality of Life based on the IBDQ questionnaire score at Week 10 and Week 20
The number of subjects with adverse events | From screening up to 2 weeks after last dose
  To evaluate the safety and tolerability of GLPG0634 in comparison with placebo in terms of adverse events (AEs)
The number of subjects with abnormal lab tests | From screening up to 2 weeks after last dose
  To evaluate the safety and tolerability of GLPG0634 in comparison with placebo in terms laboratory test abnormalities
The number of subjects with abnormal vital signs | From screening up to 2 weeks after last dose
  To evaluate the safety and tolerability of GLPG0634 in comparison with placebo in terms of abnormalities in vital signs
The number of subjects with abnormal ECG | From screening up to 2 weeks after last dose
  To evaluate the safety and tolerability of GLPG0634 in comparison with placebo in terms of abnormalities in electrocardiogram (ECG)
The plasma levels of GLPG0634 and its metabolite | Up to Week 20
  To characterize the pharmacokinetics (PK) of GLPG0634 and its metabolite by measuring the amount in plasma from Week 2 up to Week 20 at every visit
The change versus Baseline in levels of immune- and inflammation-related parameters in whole blood and serum | Up to Week 20
  To characterize the pharmacodynamics (PD) of GLPG0634 and its metabolite by measuring the levels of immune- and inflammation-related parameters in whole blood and serum
The change versus Baseline in levels of faecal calprotectin | Up to Week 20
  To characterize the pharmacodynamics (PD) of GLPG0634 and its metabolite by measuring the levels of faecal calprotectin
The change versus Baseline in microbial communities in stool samples | Up to Week 10
  To characterize the effects of GLPG0634 and its metabolite on the microbial communities by measuring the levels of predominant microbiota in stool samples

CONTACTS AND LOCATIONS:
Overall Officials: Pille Harrison, MD, Study Director — Galapagos NV
Locations (63):
- Belgium (6):
  - St. Pierre University Hospital Center, Brussels
  - University Hospital Saint Luc, Brussels
  - University Hospital Ghent, Ghent
  - University Hospitals Leuven, Leuven
  - CHR de la Citadelle, Liège
  - Clinic Saint Joseph, Liège
- Czechia (6):
  - Hepato-Gastroenterology HK Ltd., Hradec Králové
  - University Hospital Olomouc, Olomouc
  - Outpatient Clinic of Internal Medicine and Gastroenterology, Pilsen
  - Institute of Clinical and Experimental Medicine, Prague
  - Masaryk's Hospital Usti Nad Labem, Ústí nad Labem
  - Hospital Znojmo, Znojmo
- France (8):
  - Hospital Gabriel Montpied, Clermont-Ferrand
  - Beaujon Hospital, Clichy
  - Dijon University Hospital Center, Dijon
  - Hospital Michallon, Grenoble
  - Lille Regional University Hospital Center, Lille
  - North Hospital, Marseille
  - Archet Hospital, Nice
  - Saint Etienne University Hospital Center, Saint-Etienne
- Germany (8):
  - DRK Clinics Berlin Westend, Berlin
  - Interdisciplinary Crohn Colitis Center Rhein Main, Frankfurt am Main
  - Asklepios West Hospital Hamburg, Hamburg
  - University Hospital Jena, Jena
  - University Hospital Schleswig-Holstein, Kiel
  - University Hospital Magdeburg, Magdeburg
  - Gastroenterology Group Practice Minden, Minden
  - Internal Medicine Group Practice Oldenburg, Oldenburg
- Hungary (7):
  - Drug Research Center Ltd., Balatonfüred
  - Clinexpert Medical Center, Budapest
  - Semmelweis University, Budapest
  - Szent Margit Hospital, Budapest
  - University of Debrecen, Medical and Health Science Center, Debrecen
  - Bekes County Pandy Kalman Hospital, Gyula
  - Tolna County Balassa Janos Hospital, Szekszárd
- Poland (7):
  - Jan Biziel University Hospital #2, Bydgoszcz
  - Saint Family Hospital Medical Center, Lodz
  - H-T. Medical Center, Tychy
  - Clinical Hospital of Ministry of Internal Affairs and Administration, Warsaw
  - Maternal, Pediatric and Adolescent Healtcare Centre, Gastroenterology Diagnostic Facility for Adults, Warsaw
  - Vivamed, Warsaw
  - Active Health Center, Wroclaw
- Romania (4):
  - Colentina Clinical Hospital, Bucharest
  - Fundeni Clinical Institute, Bucharest
  - Medical Center for Gastroenterology, Cluj-Napoca
  - Center for Gastroenterology, Ltd, Timișoara
- Russia (13):
  - Territorial Clinical Hospital, Barnaul
  - State Medical University, Kazan'
  - Territorial Clinical Hospital, Krasnoyarsk
  - A.N. Ryzhikh State Research Center for Coloproctology, Moscow
  - City Clinical Hospital #24, Moscow
  - Moscow Clinical Research Center, Moscow
  - Vladimirsky Regional Clinical Research Institute, Moscow
  - Semashko Nizhny Novgorod Regional Clinical Hospital, Nizhny Novgorod
  - City Clinical Hospital #12, Novosibirsk
  - City Clinical Hospital #31, Saint Petersburg
  - First Pavlov State Medical University, Saint Petersburg
  - Mechnikov North-Western State Medical University, Saint Petersburg
  - St. Elizabeth City Hospital, Saint Petersburg
- United Kingdom (4):
  - Queen Elizabeth Hospital, Birmingham
  - Royal Bournemouth Hospital, Bournemouth
  - St Mark's Hospital, Harrow
  - Manchester Royal Infirmary, Manchester

REFERENCES:
- [Derived] Reinisch W, Serone A, Hebuterne X, Kuhbacher T, Klopocka M, Roblin X, Brodbeck J, Etchevers K, Galien R, Grant E, Tasset C, Yoon OK, Zaboli S, Vermeire S. Mucosal p-STAT1/3 correlates with histologic disease activity in Crohn's disease and is responsive to filgotinib. Tissue Barriers. 2023 Apr 3;11(2):2088961. doi: 10.1080/21688370.2022.2088961. Epub 2022 Jun 28. PMID 35762272
- [Derived] Vermeire S, Schreiber S, Petryka R, Kuehbacher T, Hebuterne X, Roblin X, Klopocka M, Goldis A, Wisniewska-Jarosinska M, Baranovsky A, Sike R, Stoyanova K, Tasset C, Van der Aa A, Harrison P. Clinical remission in patients with moderate-to-severe Crohn's disease treated with filgotinib (the FITZROY study): results from a phase 2, double-blind, randomised, placebo-controlled trial. Lancet. 2017 Jan 21;389(10066):266-275. doi: 10.1016/S0140-6736(16)32537-5. Epub 2016 Dec 15. PMID 27988142